CLINICAL TRIAL: NCT02061137
Title: A Phase 1 Clinical Study to Assess Safety and Efficacy of Oral Fingolimod (FTY720) in Children With Rett Syndrome.
Brief Title: Study to Assess Safety and Efficacy of Fingolimod in Children With Rett Syndrome
Acronym: FINGORETT
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University Hospital, Basel, Switzerland (Other)
Collaborators: Novartis (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CFTY720D2201T
Record Dates: First submitted 2013-08-27; First posted 2014-02-12 (Estimated); Last update posted 2018-06-15 (Actual); Status verified 2018-06

CONDITIONS: Rett's Syndrome
Keywords: Rett Syndrome (Mecp2 positive); Fingolimod (FTY 720); BDNF; Brain Atrophy
MeSH Terms: conditions — Rett Syndrome | interventions — Fingolimod Hydrochloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Rett syndrome, fingolimod (FTY720) (Experimental): 0.5 or 0.25mg Fingolimod daily
  Interventions: Drug: fingolimod (FTY720)

INTERVENTIONS:
Drug: fingolimod (FTY720) — 0.5 or 0.25 mg fingolimod orally daily for each of 6 patients with rett syndrome for 12 months
  Other Names: gilenya, fingolimod, FTY720

SUMMARY:
The Trial Objective is to assess safety and efficacy of oral fingolimod (FTY720) in children older than 6 years with Rett Syndrome. So far there is no established treatment for children with Rett Syndrome. Therefore a positive result in terms of safety and first indications of efficacy would path the way to a phase II clinical study with more patients to further test the hypothesis that fingolimod treatment may slow down the regression of motor and language skills.

DETAILED DESCRIPTION:
Rett syndrome is a neurodevelopmental disorder characterized by normal early psychomotor development followed by the loss of psychomotor and acquired purposeful hand skills and the onset of stereotyped movement of the hands and gait disturbance. The gene was discovered in 1999 and the disease was found to be caused by a mutation of the methyl-CpGbinding protein 2 (MeCP2). However, in many ways this clinically peculiar condition remains a mystery, with no clear correlations between the gene mutation and abnormal biological markers, neuropathology and/or unique clinical symptoms and signs.

Rett syndrome is an X-linked (Xq28) dominant postnatal severe neurodevelopmental disorder which is the second most common cause for genetic mental retardation in girls and the first pervasive disorder with a known genetic basis. Its incidence is between 1/10,000-15000 live births. The classical variant is characterized by apparently normal development for the first 6-18 months accompanied usually with early deceleration of head growth, followed by period of regression of motor and language skills, hand stereotypes, seizures, autonomic dysfunction and other neurological and related symptoms.

Repeated observations and experiments of the mouse models in several laboratories led to the appreciation of the role of BDNF in the disease pathophysiology. BDNF is a neurotrophic factor playing a major role in neurogenesis, neuronal survival, differentiation, and maturation during early development as well as in synaptic function and plasticity throughout life. Abnormalities in BDNF homeostasis are believed to contribute to the neurological phenotype and pathophysiology in part of the symptoms in methyl-CpG binding protein 2(Mecp2) null mice that show progressive deficits in its expression during the symptomatic stage.

FTY720 (Gilenya) is an orally active modulator of four of the five sphingosine-1 phosphate(S1P) receptors. FTY720 acts as 'super agonist' on the S1P receptor on thymocytes and lymphocytes, inducing uncoupling/internalization of that receptor.

A local study group (Yves-Alain Barde) found that FTY720 increases the levels of brain derived neurotrophic factor and improves symptoms of mice lacking MeCP2. In addition the volume of the striatum seemed to be higher (4 week old mice were treated in 4 days intervals with 0.1mg/kg body weight intraperitoneally).

Based on these results we intend to perform a phase I clinical,study to assess safety and efficacy of oral fingolimod (FTY720) in children with Rett Syndrome. Children will be included if being older than 6 years of age, fulfilling diagnostic criteria of Rett Syndrome in clinical Stages II -IV and having parents that do agree.

ELIGIBILITY:
Inclusion Criteria:

* Children fulfilling diagnostic criteria (2001, Hagberg B et al. Eur. J. Paediatr. Neurol. 2002) of Rett Syndrome
* Stages II -IV Hagberg/ Witt-Engerström (Hagberg B, Witt-Engerström I. Am J Med Genet 1986, Hagberg B. Ment Retard Dev Disabil Res Rev 2002)
* Patients older than 6 years old (have had their 6th birthday)
* Written informed consent of parents/ of legal guardian
* Negative testing for pregnancy
* Positive confirmation of a MECP2 mutation

Exclusion Criteria:

* Any uncertainty about diagnosis of Rett Syndrome
* Patients younger than 6 years old (have not yet had their 6thbirthday)
* Additional associated neurological diseases such as a brain malformation
* Patient <15kg body weight at timepoint of screening
* Patients with negative varicella-zoster virus immunoglobulin G (IgG) antibodies
* Pregnancy or breastfeeding for girls in childbearing potential age

Min Age: 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2013-08; Primary Completion 2018-04 (Actual); Study Completion 2018-04 (Actual)

PRIMARY OUTCOMES:
Levels of Brain derived neurotrophic factor (BDNF) in blood and cerebrospinal fluid before and under treatment | change of BDNF measured at Baseline, at first dose, at 6 and at 12 months after start of treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Ludwig Kappos, Prof., Principal Investigator — Department of Neurology - University Hospital Basel - Switzerland
Locations (1):
- Department of Neuropediatrics - University Children's Hospital, Basel, Switzerland

REFERENCES:
- [Derived] Naegelin Y, Kuhle J, Schadelin S, Datta AN, Magon S, Amann M, Barro C, Ramelli GP, Heesom K, Barde YA, Weber P, Kappos L. Fingolimod in children with Rett syndrome: the FINGORETT study. Orphanet J Rare Dis. 2021 Jan 6;16(1):19. doi: 10.1186/s13023-020-01655-7. PMID 33407685